CLINICAL TRIAL: NCT05457114
Title: Association Between the Use of Pulmonary Artery Catheter and Clinical Outcomes After Liver Transplantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Won Ho Kim, MD, Professor, Seoul National University Hospital
Other Study IDs: H-2205-117-1327
Record Dates: First submitted 2022-07-09; First posted 2022-07-13 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: End Stage Liver DIsease; Liver Transplant; Complications; Liver Cirrhosis; Liver Diseases
MeSH Terms: conditions — End Stage Liver Disease; Liver Cirrhosis; Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pulmonary artery catheter group: Patients who received pulmonary artery catheter insertion and hemodynamic monitoring by PAC-derived parameters
  Interventions: Device: Pulmonary artery catheter (Edward Lifesciences, Irvine, California, USA)
- Non-pulmonary artery catheter group: Patients who did not received pulmonary artery catheter insertion and were monitored with Flo-Trac FloTrac Vigileo
  Interventions: Device: FloTrac Vigileo system (EV1000 clinical platform, Edward Lifesciences, Irvine, California, USA)

INTERVENTIONS:
Device: Pulmonary artery catheter (Edward Lifesciences, Irvine, California, USA) — PAC was inserted and connected to a continuous cardiac output monitor (Vigilance I from 2006 to 2012; Vigilance II from 2012 to 2022, Edward Lifesciences, Irvine, USA)
  Groups: Pulmonary artery catheter group
Device: FloTrac Vigileo system (EV1000 clinical platform, Edward Lifesciences, Irvine, California, USA) — Without PAC, monitoring with FloTrac Vigileo system (EV1000 clinical platform, Edward Lifesciences, Irvine, California, USA) was performed for continuous cardiac output monitoring.
  Groups: Non-pulmonary artery catheter group

SUMMARY:
The investigators attempted to evaluate whether the use of PAC is associated with better clinical outcomes after liver transplantation compared with the case without PAC.

DETAILED DESCRIPTION:
Pulmonary artery catheter (PAC) has been used for advanced hemodynamic monitoring during liver transplantation. However, recent advances in less invasive monitoring could provide continuous cardiac output monitoring by arterial waveform analysis. Using this technology, stroke volume variation (SVV) is monitored as a preload index. Calculated systemic vascular resistance (SVR) can be monitored if central venous pressure (CVP) is provided. Therefore, this less invasive form of hemodynamic monitoring may replace the PAC. The investigators attempted to evaluate whether the use of PAC is associated with better clinical outcomes after liver transplantation compared with the case without PAC.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who underwent living or deceased donor liver transplantation at our tertiary care university hospital between 2006 and 2022

Exclusion Criteria:

* Patients with baseline renal dysfunction
* Missing baseline or outcome variables
* Retransplantation
* Patients who received intraoperative transesophageal echocardiography (TEE) monitoring

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients received liver transplantation surgery in a single tertiary care university hospital
Sampling Method: Non-Probability Sample
Enrollment: 1970 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with acute kidney injury | the first 7 postoperative days
  Acute kidney injury (AKI) was defined by the Kidney Disease Improving Global Outcomes (KDIGO) criteria, which was defined according to the greatest change in serum creatinine level during the postoperative seven days (Stage 1: more than 1.5-fold; stage 2: more than 2-fold; stage 3: more than 3-fold increase from baseline level or increase in serum creatinine to ≥ 4.0 mg/dL or the initiation of renal replacement therapy). The most recent serum creatinine level measured before surgery was collected as a baseline value.
Number of Participants with early allograft dysfunction | the first 7 postoperative days
  Early allograft dysfunction (EAD) was defined when one or more of the following are present within the first 7 postoperative days: total bilirubin ≥ 10 mg/dL, prothrombin time: international normalized ratio ≥ 1.6, or aspartate or alanine transaminase > 2000 IU/L

SECONDARY OUTCOMES:
In-hospital mortality | the first month after admission
  all-cause mortality during hospitalization
One-year mortality | one year after transplantation
  all-cause mortality during one year after transplantation
Length of intensive care unit (ICU) stay | the first month after admission
  Length of intensive care unit stay after transplantation
Length of hospital stay | the first month after admission
  Length of hospital stay after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Won Ho Kim, MD, PhD, Study Chair — Department of Anaesthesiology and Pain Medicine, Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jung JY, Sohn JY, Lim L, Cho H, Ju JW, Yoon HK, Yang SM, Lee HJ, Kim WH. Pulmonary artery catheter monitoring versus arterial waveform-based monitoring during liver transplantation: a retrospective cohort study. Sci Rep. 2023 Nov 15;13(1):19947. doi: 10.1038/s41598-023-46173-1. PMID 37968287